CLINICAL TRIAL: NCT01548196
Title: A Prospective, Randomized Controlled Pilot Study Of Standard Percutaneous Nephrolithotomy (PNL) Versus Tubeless PNL Versus Tubeless Stentless PNL
Brief Title: Standard Percutaneous Nephrolithotomy Percutaneous Nephrolithotomy (PNL) Versus Tubeless PNL Versus Tubeless Stentless PNL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00004138
Record Dates: First submitted 2011-10-18; First posted 2012-03-08 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2012-03

CONDITIONS: Nephrolithotomy
Keywords: nephrolithotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- standard percutaneous nephrostomy (Other): Standard PCN
  Interventions: Procedure: Standard Percutaneous nephrolithotomy
- double-J ureteral stent, (Other): double-J ureteral stent,
  Interventions: Procedure: Standard Percutaneous nephrolithotomy
- open-ended ureteral catheter (Other): open-ended ureteral catheter
  Interventions: Procedure: Standard Percutaneous nephrolithotomy
- no nephrostomy or ureteral stent/catheter. (No Intervention): no nephrostomy or ureteral stent/catheter.

INTERVENTIONS:
Procedure: Standard Percutaneous nephrolithotomy — Percutaneous nephrolithotomy
  Arms: double-J ureteral stent,; open-ended ureteral catheter; standard percutaneous nephrostomy

SUMMARY:
The purpose of the study is to assess and compare the efficacy and morbidity standard percutaneous nephrolithotomy with tubeless PNL. A total of approximately 60 patients will be enrolled. Patients will be randomized to one of four groups: standard percutaneous nephrostomy, double-J ureteral stent, open-ended ureteral catheter and no nephrostomy or ureteral stent/catheter. Primary Outcome Measures will include length of procedure and estimated blood loss. Post-operative analgesic use (both parenteral and oral), pain scores, time to ambulation, time to oral intake, and pain scores will also be recorded. Time to nephrostomy tube removal, external ureteral and Foley catheter removal and patient discharge from the hospital will also be recorded. Incidence and type of post-operative complications will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Planned single tract percutaneous nephrolithotomy
* General anesthesia for percutaneous nephrolithotomy

Exclusion Criteria:

* Age<18 years old
* Known residual calculi at the end of the procedure
* Significant hemorrhage during procedure
* Bleeding disorder (This does not include patients taking anti-coagulants as these are stopped prior to surgery.)
* Prisoners
* Inability to give informed consent
* Pregnant females
* Solitary kidney
* Transplant kidney
* Pleural effusion during procedure requiring drainage
* Perforation of renal collecting system during procedure
* Incomplete stone clearance
* Chronic pain syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | until hospital discharge, about 2-3 days
  measuring days of hospital stay after procedure, and the effect that the location of the puncture has on the length of hospital stay
Change in CBC and Chemistry Panel | at time of hospital discharge, about 2-3 days
  Loss of blood

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Preminger, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States